CLINICAL TRIAL: NCT04874753
Title: The Effect of COVID-19 Pandemia on Follow up of Patients With Chronic Kidney Disease
Acronym: COVID19-CKD
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Zelal Adibelli, Assistant Prof. Zelal Adibelli, Uşak University
Other Study IDs: UsakU4
Record Dates: First submitted 2021-05-02; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Chronic Kidney Diseases; Proteinuria
MeSH Terms: conditions — COVID-19; Renal Insufficiency, Chronic; Proteinuria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: change in kidney function and proteinuria — change in eGFR nad proteinuria in patients with chronic kidney disease

SUMMARY:
COVID-19 pandemic affected the admission of patients to the hospital especially the older patients (> 65 years old) because of curfews and the reluctance of patients to apply to the hospitals. Chronic kidney disease is characterized with the progressive loss of kidney function over the time and regular follow-up of patients for their kidney function and treatment of complications is recommended in these patients.

DETAILED DESCRIPTION:
The chronis kidney disease patients followed in Nephrology outpatient unit are going to be enrolled in the study and their kidney functions (calculated with the mdrd formula to asses the estimated glomerular filtration rate (eGFR)) will be evaluated 6 months before and after the COVID-19 pandemia. And the rate of initiation of renal replacement therapies and the change in proteinuria will be evaluated 6 months before and after the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic kidney disease on regular follow-up for 6 months before the COVID19 pandemic.

Exclusion Criteria:

* patients without chronic kidney disease
* patients not on routine follow-up for 6 months before the COVID19 pandemic

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic kidney disease (eGFR<60 ml/dk) between the ages 18-80 followed up in nephrology outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
eGFR change | 6 months
  a rise or decrease in eGFR
change in proteinuria | 6 months
  increase or decrease in ptoteinuria levels

SECONDARY OUTCOMES:
initiation of renal replacement therapies | 6 months
  need for hemodialysis or peritoneal dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Zelal Adıbelli, Principal Investigator — Uşak University
Locations (1):
- Usak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided